CLINICAL TRIAL: NCT01929122
Title: BENEFIT: Beans/Bran Enriching Nutritional Eating For Intestinal Health Trial
Brief Title: Beans/Bran Enriching Nutritional Eating For Intestinal Health Trial
Acronym: BENEFIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Poudre Valley Health System (Other)
Responsible Party: Principal Investigator, Elizabeth P Ryan, Assistant Professor of Toxicology and Nutrition, Colorado State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 10-1038; 1R21CA161472-01A1 (NIH)
Record Dates: First submitted 2013-08-22; First posted 2013-08-27 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Colorectal Cancer Control and Prevention
Keywords: Prevention & control; Diet; Functional food; Nutrition Assessment; Oryza sativa; Rice Bran; Phaseolus vulgaris L.; Legumes; Microbiome; Metabolomics; Prebiotics
MeSH Terms: interventions — Snacks

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo-Control (Placebo Comparator): Randomized participants consume 1 meal and 1 snack per day that does not include either rice bran or navy bean powder for 28 days.
  Interventions: Dietary Supplement: Placebo-Control Meals and Snacks
- Cooked Navy Bean Powder (Experimental): Randomized participants consume 1 meal and 1 snack per day containing cooked navy bean powder (35 g/day) for 28 days.
  Interventions: Dietary Supplement: Cooked Navy Bean Powder Meals and Snacks
- Rice Bran (Experimental): Randomized participants consume 1 meal and 1 snack per day containing rice bran (30 g/day) for 28 days.
  Interventions: Dietary Supplement: Rice Bran Meals and Snacks

INTERVENTIONS:
Dietary Supplement: Placebo-Control Meals and Snacks
  Other Names: Whole food dietary intervention
  Arms: Placebo-Control
Dietary Supplement: Cooked Navy Bean Powder Meals and Snacks
  Other Names: Whole food dietary intervention
  Arms: Cooked Navy Bean Powder
Dietary Supplement: Rice Bran Meals and Snacks
  Other Names: Whole food dietary intervention
  Arms: Rice Bran

SUMMARY:
The purpose of this study is to explore the effects of cooked navy bean powder or rice bran consumption on the stool microbiome and metabolome of colorectal cancer survivors and healthy adults.

DETAILED DESCRIPTION:
Objectives:

1. To learn about how increased cooked navy bean powders or rice bran dietary intake affect the stool microbiota of colorectal cancer survivors and healthy adults.
2. To determine whether cooked navy bean powders or rice bran consumption modulate microbial metabolism.
3. To observe dietary changes in the blood, urine and stool metabolite profiles and inflammatory cytokines.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age.
* Be a Colorectal Cancer Survivor that is a minimum of 4 months post chemotherapy/radiation treatment. OR be a healthy adult with no prior history of treatment for cancer.
* BMI between 25-35
* no previous or concurrent malignancy except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer and other cancer for which the patient has been disease free for five years.
* Ability to complete questionnaire(s) and dietary food logs
* Willingness to consume meals/snacks provided for 28 consecutive days
* Drink less than or equal to one alcoholic drink/day

Exclusion Criteria:

* History of food allergies and/or major dietary restrictions
* Pregnant or lactating or planning to become pregnant
* Self identified as a smoker
* Taking prescribed medication to control their lipids
* Taking Bean-O, other anti-flatulence medications or prolonged antibiotic use (one month)
* Have a history of gallstones.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2010-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Stool Microbiome Composition and Metabolome | 5 years

SECONDARY OUTCOMES:
Navy Bean or Rice Bran metabolites in stool, urine and blood. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth P Ryan, PhD, Principal Investigator — Colorado State University
Locations (2):
- United States (2):
  - Colorado State University, Fort Collins, Colorado
  - Poudre Valley Hospital Oncology Research, Fort Collins, Colorado

REFERENCES:
- [Result] Borresen EC, Gundlach KA, Wdowik M, Rao S, Brown RJ, Ryan EP. Feasibility of Increased Navy Bean Powder Consumption for Primary and Secondary Colorectal Cancer Prevention. Curr Nutr Food Sci. 2014 May;10(2):112-119. doi: 10.2174/1573401310666140306005934. PMID 25009453
- [Result] Borresen EC, Brown DG, Harbison G, Taylor L, Fairbanks A, O'Malia J, Bazan M, Rao S, Bailey SM, Wdowik M, Weir TL, Brown RJ, Ryan EP. A Randomized Controlled Trial to Increase Navy Bean or Rice Bran Consumption in Colorectal Cancer Survivors. Nutr Cancer. 2016 Nov-Dec;68(8):1269-1280. doi: 10.1080/01635581.2016.1224370. Epub 2016 Sep 30. PMID 27689688
- [Result] Sheflin AM, Borresen EC, Kirkwood JS, Boot CM, Whitney AK, Lu S, Brown RJ, Broeckling CD, Ryan EP, Weir TL. Dietary supplementation with rice bran or navy bean alters gut bacterial metabolism in colorectal cancer survivors. Mol Nutr Food Res. 2017 Jan;61(1):10.1002/mnfr.201500905. doi: 10.1002/mnfr.201500905. Epub 2016 Sep 12. PMID 27461523
- See also: Related Information — http://csu-cvmbs.colostate.edu/academics/erhs/Pages/elizabeth-ryan-lab-human-studies.aspx